CLINICAL TRIAL: NCT04627246
Title: A Phase Ib Study of the Combination of Personalized Autologous Dendritic Cell Vaccine and Standard of Care Adjuvant Chemotherapy Followed by Nivolumab for Resected Pancreatic Adenocarcinoma
Brief Title: Personalized Vaccine with SOC Chemo Followed by Nivo in Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Antonia Digklia, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-0011-PC_PEP-DC_2017
Record Dates: First submitted 2020-10-15; First posted 2020-11-13 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreas; vaccine; nivolumab; cancer; adenocarcinoma
MeSH Terms: conditions — Neoplasms; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: A total of 12 evaluable patients will be recruited. They will receive the same investigational products.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEP-DC + Nivolumab + SOC (Experimental): PEP-DC: Autologous Dendritic Cell Vaccine Loaded with Personalized Peptides Nivolumab SOC: Standard of Care Chemotherapy
  Interventions: Biological: Autologous Dendritic Cell Vaccine Loaded with Personalized Peptides (PEP-DC vaccine)

INTERVENTIONS:
Biological: Autologous Dendritic Cell Vaccine Loaded with Personalized Peptides (PEP-DC vaccine) — SOC: Subgroup1: intravenous mFOLFIRINOX for twelve 14-day cycles. Subgroup2: intravenous gemcitabine twice, on days 1 and 8, and oral capecitabine for 14 days of 21-day cycles, for eight cycles.
  PEP-DC vaccine: At least 5 subcutaneous vaccinations starting on cycle 8 (subgroup1) or cycle 5 (subgroup2) of chemotherapy: Subgroup1: every 4 weeks, on day 3 of every second 14-day cycle, and then every 4 weeks starting from the first nivolumab administration. Subgroup2: Every 3 weeks, on day 9 of each 21-day cycle, and then every 4 weeks starting from the second nivolumab administration.
  Nivolumab for a maximal duration of 2 years: intravenous, starting after the last chemotherapy cycle. Administered as flat dose of 240mg every 2 weeks during 14 weeks, then as flat dose of 480 mg every 4 weeks until the last vaccination. Then, as a maintenance therapy at 480 mg every 4 weeks until appearance of new lesions or unacceptable toxicity.

SUMMARY:
Phase Ib clinical trial using Autologous Dendritic Cell Vaccine Loaded with Personalized Peptides (PEP) in order to stimulate/induce both innate and adaptive immunity by activating T-cells and Natural Killer (NK) cells, combined with standard of care (SOC) adjuvant chemotherapy, followed by nivolumab, an antibody against Programmed Cell Death 1 (PD-1), to maintain and boost the vaccine's effect in patients with non-metastatic resectable pancreatic adenocarcinoma

DETAILED DESCRIPTION:
This is a single center, single arm, phase Ib trial to evaluate the feasibility, safety, immunogenicity, and efficacy of subcutaneous dendritic cell (DC) vaccine loaded with personalized peptides [PEP-DC vaccine] in combination with standard of care adjuvant chemotherapy (subgroup 1: mFOLFIRINOX or subgroup 2: gemcitabine and capecitabine), followed by the antibody nivolumab in patients with non-metastatic surgically resected pancreatic adenocarcinoma.

All patients will have previously undergone collection of resected advanced pancreatic tumor tissue under a different research protocol with a separate informed consent. After registration, all patients will receive standard of care chemotherapy:

Subgroup 1: intravenous mFOLFIRINOX for twelve 2-week cycles. Subgroup 2: intravenous gemcitabine, and oral capecitabine for eight 21-day cycles. Additionally, all eligible patients will undergo apheresis during the cycle 5 of mFOLFIRINOX (subgroup 1) or the last week of cycle 3 of gemcitabine/ capecitabine (subgroup 2) to collect peripheral blood mononuclear cells (PBMCs) for dendritic cell vaccine production. All patients will receive at least six PEP-DC vaccinations starting concomitant with the 8th cycle (subgroup 1) or the 5th cycle (subgroup 2) of chemotherapy.

Subgroup 1: Vaccine will be delivered subcutaneously every 4 weeks, on day 3(+1) of every second 14-day cycle, and thereafter every four weeks starting from the first nivolumab administration.

Subgroup 2: Vaccine will be administered subcutaneously every 3 weeks, on day 9 (the day after last gemcitabine infusion) of each 21-day cycle, and thereafter every four weeks starting from the second nivolumab administration.

Nivolumab will be administered intravenously over a period of 30 minutes to all patients, for a maximum duration of 2 years, as follows:

Subgroup 1: Nivolumab treatment will start after the last cycle of chemotherapy (2 weeks after C12D1) and will be given as flat dose of 240 mg given every 2 weeks, during 14 weeks (2-week cycles). Then it will be administered as flat dose of 480 mg every 4 weeks (4-week-cycles), until the last vaccine dose.

Subgroup 2: Nivolumab treatment will start after the last cycle of chemotherapy (3 weeks after C8D1) as flat dose of 240 mg given every 2 weeks, for 14 weeks. Then it will be administered as flat dose of 480 mg every 4 weeks, until the last vaccine dose. Nivolumab treatment should be maintained for at least for 8 weeks after end of the last chemotherapy cycle if vaccination stops earlier.

Nivolumab maintenance for both subgroups: After the end of combined treatment period (vaccination plus nivolumab), nivolumab will be given at 480 mg (flat dose) every four weeks to all patients until appearance of new lesions, unacceptable toxicity or until the maximum time for nivolumab treatment (2 year) is reached.

Regular physical examination, radiological evaluation and blood testing for safety parameters will be performed according to the schedule during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Histologically confirmed resected adenocarcinoma of the pancreas (T1-T4, N 0-1-2, minimum 2cm - American Joint Committee on Cancer (AJCC) 8th edition).

  * Mixed adenocarcinoma tumors are eligible provided the predominant invasive component of the tumor is adenocarcinoma
  * Patients who received or did not receive neo-adjuvant chemotherapy are eligible, both.
* No distant metastasis
* Appropriate amount of tumoral tissue was collected from the cytoreductive surgery and allowed the identification of top 10 personalized peptides (PEP) for preparation of PEP-DC vaccine
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Adequate hematologic and end-organ function, defined by the following laboratory results obtained within 21 days prior registration
* Adequate serology defined by the following laboratory results:

  * Negative test for human immunodeficiency viruses (HIV)
  * Patients with active or chronic hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at pre-screening) are not eligible.
  * Patients with past/resolved hepatitis B virus (HBV) infection (defined as having a negative hepatitis B surface antigen (HBsAg) test and a positive antibody to hepatitis B core antigen (anti-HBc) antibody test) are eligible, if hepatitis B virus deoxyribonucleic acid (HBV DNA) test is negative.
  * Hepatitis B virus deoxyribonucleic acid (HBV DNA) must be obtained in patients with positive hepatitis B core antibody prior start of study treatment.
  * Patients with active hepatitis C are not eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if Polymerase Chain Reaction (PCR) is negative for hepatitis C virus ribonucleic acid (HCV RNA)
* No measurable tumor lesion according to radiologic criteria (New Response Evaluation Criteria in Solid Tumours 1.1 (RECIST 1.1))
* Recovery from any toxic effects of prior neo-adjuvant therapy to less than Grade 1 per the National Cancer Institute Common Terminology Criteria for Adverse Events v4.03 except for toxicities described below, as long as they do not put at risk the patient's condition and do not require systemic immunosuppressive steroids at any dose, including but not limited to:

  * Fatigue
  * Alopecia
  * Skin disorders
  * Stable neuropathy
  * Endocrinopathies requiring replacement treatment

Note: For other medical conditions, or for any other toxicity with a higher grade but controlled by adequate treatment, prior discussion and agreement with the principal investigator is mandatory.

Note: Patients may have undergone surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.

* For women of childbearing potential (sexually mature women who have not undergone a hysterectomy, have not been naturally post-menopausal for at least 12 consecutive months or have a serum follicle-stimulating hormone (FSH) less than 40 milli international unit per milliliter (mIU/ml):

  1. Agreement to follow instructions for methods of contraception for the couple from screening until 6 months after last vaccine dose, or last chemotherapy treatment, or last nivolumab treatment
  2. Women of childbearing potentia must have a negative urine pregnancy test within 7 days, before registration. A positive urine test must be confirmed by a serum pregnancy test.
* For men and their female partners: agreement to follow instructions for methods of contraception for the couple from screening until 7 months after last vaccine dose, or last chemotherapy treatment, or last nivolumab treatment.
* Patient is able to undergo leukapheresis

Exclusion Criteria:

* Pregnant or breast-feeding women
* Other malignancy within 2 years prior study enrollment, except for those treated with surgical intervention as curative intent. Patients with a predicted 5-year recurrence-free survival rate equal or more than 95% can be included at the investigator's discretion.
* Current, recent (within 4 weeks prior registration), or planned participation in an experimental drug study.
* Past history with cardiac problem:

  * New York Heart Association Class II or greater congestive heart failure
  * History of myocardial infarction or unstable angina within 6 months prior registration. History of stroke or transient ischemic attack within 6 months prior registration.
  * Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior registration.
  * Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Known hypersensitivity to any component of the study treatment
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

The following exceptions are considered:

* Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study.
* Patients with controlled Type I diabetes mellitus on a stable insulin regimen are eligible
* Psoriasis not requiring systemic treatment.
* Vitiligo.
* Other conditions not expected to recur in the absence of an external trigger, are permitted to enroll after agreement with the principal investigator.

  - Severe infections within 8 weeks prior registration including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia or signs or symptoms of infection requiring oral or intravenous antibiotics within 8 weeks prior registration.
* Patients receiving routine antibiotic prophylaxis (e.g., to prevent chronic obstructive pulmonary disease exacerbation or for dental extraction) are eligible.

  - Administration of a live, attenuated vaccine within 8 weeks before registration
* Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine within 4 weeks prior registration or at any time during the study.

  * Dihydropyrimidine dehydrogenase deficiency
  * Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
  * Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may impair the ability of the subject to receive protocol therapy and comply with study visits and procedures.
  * Patients who have received prior treatment with anti-programmed cell death 1 (PD1), anti-programmed death ligand 1 (PD-L1) or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) may be enrolled, provided at least 5 half-lives have elapsed from the last dose to the first dose of nivolumab and there was no history of severe immune-mediated adverse effects from such therapy (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 and 4).
  * Treatment with systemic immunostimulatory agents (including but not limited to interferon-alpha, interleukin-2) for any reason within 4 weeks or five half-lives of the drug, whichever is shorter, prior to registration.
  * Treatment with systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior registration.
* Patients who are receiving acute, low-dose, systemic immunosuppressant medications (e.g., an one-time dose of dexamethasone for nausea) or physiologic replacement doses (i.e., prednisone 5-7.5 mg/day, or other) for adrenal insufficiency may be enrolled in the study.
* The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.

  * Treatment with Granulocyte colony-stimulating factor within 4 weeks prior registration.
  * Treatment with K-vitamin antagonists such as warfarin unless it is switched to another type of anticoagulant treatment, if the patient is assigned to receive capecitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of cases for which vaccine is produced | 3 years after study activation
  Feasibility will be assessed measuring the number of cases, in which vaccine is produced successfully (defined as production and quality control release of at least 5 PEP-DC vaccines for a patient) among the enrolled patients and number of patients who receive at least one dose of vaccine
Assessment of adverse events | 3 years after study activation
  Collection of adverse events and serious adverse events, treatment limiting toxicities and assessment of immunogenicity

SECONDARY OUTCOMES:
Relapse free survival | 8 years
  Time from enrolment (registration) date until one of the following events: a. patients disease-free at inclusion, until first date of documented progression, b. patients with non-measurable lesions at inclusion, until first date of documented progression, c. death
Overall survival | 8 years
  Time from enrolment (registration) date to date of death due to any cause, or last patient contact. For living patients, the date of most recent clinic visit or a phone or email contact will be employed to document the overall survival time.
Gene analysis of immunological response | 8 years
  The assessment of the interactions between tumor cells and the immune system within the tumor microenvironment will be performed by gene expression quantification using with multiplex gene expression profiling.
Cell analysis of immunological response | 8 years
  The assessment of the interactions between tumor cells and the immune system within the tumor microenvironment will be performed by cell quantification using with multi-parametric single-cell cytometry and single cell RNA sequencing analysis
Evaluation of tumor marker carbohydrate antigene 19-9 (CA19-9) or carcinoembryonic antigen (CEA) kinetics | 8 years
  Measurement of tumoral markers by blood analysis
Correlation between immune-related adverse events and relapse-free survival | 8 years
  Number of immune-related adverse events using the CTCAE v.4.03 correlated with relapse-free survival (time in months)

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV Oncology Department, Lausanne, Canton of Vaud, Switzerland